CLINICAL TRIAL: NCT05090631
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: The Role of Genetic Factors in the Development of Atopic Dermatitis in the Kazakh Population
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1196
Record Dates: First submitted 2021-09-25; First posted 2021-10-25 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis
Keywords: GWAS
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: Patients with atopic dermatitis
  Interventions: Genetic: DNA analysis
- Control group: Patients without atopic dermatitis
  Interventions: Genetic: DNA analysis

INTERVENTIONS:
Genetic: DNA analysis — GWAS

SUMMARY:
This is a GWAS study that aims to identify possible candidate genes associate to atopic dermatitisby exploring single nucleotide polymorphism (SNP) in a group of atopic dermatitis, in the Kazakh population. The investigators hypothesize that the careful phenotyping of the subject sand matching with increase the power to find SNP significantly associate with atopic dermatitis

DETAILED DESCRIPTION:
A genome-wide association study (GWAS) is an approach used in genetics research to associate specific genetic variations with particular diseases. The method involves scanning the genomes from many different people and looking for genetic markers that can be used to predict the presence of a disease. Once such genetic markers are identified, they can be used to understand how genes contribute to the disease and develop better prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Persons with various forms of a confirmed diagnosis of atopic dermatitis;
* The age of the patients is from 18 to 45+ years;
* Persons of Kazakh nationality, whose paternal and maternal grandparents are Kazakhs.
* Persons who are able and willing to provide written informed consent;
* Persons capable and willing to comply with the research protocol;

Exclusion Criteria:

* Persons under the age of 18;
* Patients with severe concomitant systemic diseases, including cardiovascular, respiratory, hepatic and renal failure
* Patients with severe infectious processes (sepsis, abscess, hepatitis B and C, HIV)
* Persons with mental illness.
* Persons taking corticosteroid drugs, immunosuppressants within the last month;
* Persons who, in the opinion of the researcher, are mentally or legally incapacitated, which prevents obtaining informed consent;
* Pregnant or lactating women;
* Tuberculosis of any localization in the active phase and in history;
* Severe and decompensated diseases of the liver and kidneys, cardiovascular system;
* Severe and decompensated course of endocrine diseases;
* Autoimmune diseases;
* Systemic diseases;
* Oncological diseases;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: KAZAKH POPULATION
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-10-23 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
number of SNPs associated with atopic dermatitis | 1 year
  Using GWAS to identify candidate genes associate with atopic dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Gulya Sarybaeva, PhD, Principal Investigator — Asfendiyarov Kazakh National Medical University
Locations (1):
- Kazakhstan, Almaty, Kazakhstan